CLINICAL TRIAL: NCT03918486
Title: Caretaker vs. Routine Blood Pressure Sphygmomanometer
Status: Completed | Type: Observational
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 17-119EX
Record Dates: First submitted 2018-10-10; First posted 2019-04-17 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Caretaker: Comparing blood pressure obtained using routine blood pressure sphygmomanometer to a non-invasive device that continuously monitors central blood pressure (CareTaker).
  Interventions: Device: Caretaker

INTERVENTIONS:
Device: Caretaker — Application of Caretaker device to subjects that are scheduled for elective surgeries.

SUMMARY:
Caretaker vs. routine blood pressure sphygmomanometer

DETAILED DESCRIPTION:
The aim of this study is to: Compare blood pressure obtained using routine blood pressure sphygmomanometer to a non-invasive device that continuously monitors central blood pressure (CareTaker).

ELIGIBILITY:
Inclusion Criteria:

* Adults ages > 18 who are having their blood pressure monitored using routine blood pressure sphygmomanometer.

Exclusion Criteria:

* Patients not scheduled to be monitored using blood pressure sphygmomanometer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ages > 18 who are having their blood pressure monitored using routine blood pressure sphygmomanometer.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Comparing blood pressure using routine blood pressure cuff to that recorded by the Caretaker device. | Length of surgery
  As per blood pressure monitor validation guidelines, the primary outcome measure will be the average difference in systolic and diastolic blood pressure measurements between the investigational device (Caretaker) and the reference (brachial cuff). In line with the ANSI/ISO/AAMI guidelines, we will obtain multiple investigational-reference measurement pairs in each subject (every 5 minutes during the surgical case) and will average the difference over all pairs from all subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States